CLINICAL TRIAL: NCT00934115
Title: Epidemiology of Infections in Pediatric Cancer Patients: A Prospective Multicenter Study in Israel
Brief Title: Epidemiology of Infections in Pediatric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Itzhak Levy MD, Schneider Children Medical Center
Other Study IDs: 0061-07-RMC
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Infections
Keywords: To define the incidence, categories of infections by organ systems, etiologic agents and risk
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Infections are common causes of morbidity and mortality in pediatric cancer patients. Today, there are limited data on the incidence, distribution of specific infections, causative agents and risk factors for severe infections in this population. Moreover, little data exist on the epidemiology of infections among pediatric patients with solid tumors.

The objectives of the present study are to define the incidence, categories of infections by organ systems, etiologic agents and risk factors for infections in different pediatric malignancies. The results of this study will help the investigators to better understand the epidemiology of infections in the different types of pediatric malignancies, enable the investigators to identify high risk patients, and design a better approach to empiric treatment of these patients.

A prospective, multi-center study, conducted in 5 pediatric hematology-oncology units across Israel (Rambam Medical Center, Haemek Medical Center, Schneider Children's Medical Center, Hadassah Medical Center, Soroka Medical Center). All children aged 0-18 years of age, newly diagnosed with cancer and admitted to day care or inpatient departments with fever of >38.0 C will be included in the study. Demographic, clinical and microbiological figures will be collected in each center by a research assistant supervised by the infectious disease specialist. Data will be collected according to a pre-defined Patient Data Form and entered into an electronic data base that will be analyzed accordingly. In each event of febrile episode during chemotherapy, the following data will be collected by a research assistant using a patient data form and computerized software:

* Demographic data: age, gender, ethnicity.
* Clinical data: Underlying disease, immunizations, prophylactic antibiotics, presence of central venous catheter, intensity of chemotherapy, duration of fever, duration and severity of neutropenia, diagnosis of present event.
* Imaging data
* Microbiological data
* Outcome

The statistical analysis will be performed by an epidemiologist and statistician using the SPSS 12.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cancer patients admitted to hospital with fever

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01